CLINICAL TRIAL: NCT07193966
Title: Safety and Efficacy of NG2 and DLL3 CAR-T Therapy Targeting Melanoma
Brief Title: NG2 and DLL3 CAR-T Cells Targeting Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-25004
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: melanoma; CAR-T; chimeric antigen receptor; adoptive T cell transfer; NG2; DLL3
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effectiveness of CAR-T cells targeting NG2 and DLL3 (Experimental): Gene-modified T cells are designed to kill tumor cells through specific recognition of NG2 and DLL3. This study will evaluate the side effects and effective doses of NG2 and DLL3 CAR-T cells in treating refractory and recurrent melanoma
  Interventions: Biological: NG2 and DLL3 CAR-T cells

INTERVENTIONS:
Biological: NG2 and DLL3 CAR-T cells — Infusion of NG2 and DLL3-specific CAR-T via intravenous route

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of multiple CAR-T cell therapy which targets NG2 and DLL3 surface antigens in patients with relapsed and refractory melanoma.

DETAILED DESCRIPTION:
Melanoma, known for having the highest mutation burden among solid tumors, is in a steady rise in incidence over recent years. Early-stage melanoma can be treated by surgery. As the tumor invades deeper and cancer cells metastasize, the difficulty of radical surgery increases, and melanoma is highly resistant to conventional chemotherapy and radiation therapy. In this context, immunotherapy has become a new area of exploration.

NG2 (chondroitin sulfate protein polysaccharide 4) is a cell surface type I transmembrane proteoglycan with substantial advantages as a potential therapeutic target for melanoma. On one hand, it exhibits strong targeting specificity, showing high expression in melanoma cells and in tumor angiogenesis-related blood vessels while maintaining low expression in normal tissues. This enables its targeted delivery to tumor sites, reducing damage to healthy tissues and minimizing side effects. On the other hand, NG2 involves multiple mechanisms: it not only participates in melanoma cell proliferation and survival but also plays a crucial role in tumor angiogenesis. Targeting NG2 may simultaneously inhibit both tumor cell growth and angiogenesis. Additionally, NG2 demonstrates prognostic value, as studies show its high expression correlates with better disease-free survival (DFS) in melanoma patients. This makes it a prognostic marker that helps assess disease progression and prognosis, providing valuable insights for treatment regimen formulation.

Another potential therapeutic target, delta-like ligand 3 (DLL3), demonstrates three key advantages: first, it exhibits high targeting specificity - showing low expression in normal tissues but high expression in melanoma cells. This enables precision targeting by related drugs (such as antibody conjugates ADCs and CAR-T) to effectively attack tumors while minimizing damage to healthy tissues and reducing toxic side effects. Second, it restoring Notch signaling to inhibit tumor cell growth while blocking angiogenesis and epithelial mesenchymal transition (EMT), thereby suppressing cancer progression from both cellular and microenvironmental dimensions. Third, it shows broad clinical prospects, serving as a prognostic marker to guide personalized treatment and providing new therapeutic options for DLL3-positive patients with poor response to PD-1 inhibitors, potentially breaking through the treatment bottleneck in advanced melanoma.

The purpose of this clinical study is to assess the feasibility, safety and efficacy of the combinational NG2 and DLL3 CAR T cell immunotherapy in patients who have melanoma in relapsed state or late stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors have received standard first-line therapy and have been diagnosed with non-resectable, metastatic, progressive or recurrent conditions.
* The expression status of NG2 and DLL3 antigens of the tumor has been determined for eligibility. Positive expression is defined by NG2 and DLL3 antibody staining results based on immunohistochemistry or flow cytometry analyses.
* Body weight greater than or equal to 40 kg.
* Age: ≥18 year and ≤ 75 years of age at the time of enrollment.
* Life expectancy: at least 8 weeks.
* Prior Therapy:

  1. There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less.
  2. Participants must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection.
  3. At least 7 days must have elapsed since the completion of therapy with any biologic agent, targeted agent, tyrosine kinase inhibitor or metronomic non-myelosuppressive regimen.
  4. At least 4 weeks must have elapsed since prior therapy that includes a monoclonal antibody.
  5. At least 1 week must has elapsed since any radiation therapy at the time of study entry.
* Karnofsky/jansky score of 70% or greater.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent.
* Pulse Ox greater than or equal to 90% on room air.
* Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
* Renal function: Patients must have serum creatinine less than 3 times ULN.
* Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease not evaluable for hematologic toxicity.
* For all patients enrolled in this study, their parents or legal guardians must sign an informed consent and assent.

Exclusion Criteria:

* Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, with the exception of grade 3 hematologic toxicity.
* Untreated central nervous system (CNS) metastasis; patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
* Previous treatment with other genetically engineered CAR T cells.
* Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
* Patients who require systemic corticosteroid or other immunosuppressive therapy.
* Evidence of tumor potentially causing airway obstruction.
* Inability to comply with protocol requirements.
* Insufficient availability of CART cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 3 months
  Determine the toxicity profile the NG2 and DLL3 cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 1 year
  Disease status is defined by image scan to get the outcomes such as Complete response/remission (CR), Very good partial response/remission (VGPR), etc.
The persistence of anti-NG2 and DLL3 CAR-T cells | 1 year
  The investigators will monitor the scale of NG2 and DLL3 CAR-T cells in the peripheral blood.
Survival time of the patients | 3 year
  The survival time of the patients treated with the NG2 and DLL3 CAR-T cells will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No